CLINICAL TRIAL: NCT02571478
Title: Evaluation of a Brief Marriage Intervention for Internal Behavioral Health Consultants in Military Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wright State University (Other)
Collaborators: Clark University (Other); 59th Medical Wing (U.S. Federal Agency); Malcolm Grow Medical Clinics and Surgery Center (U.S. Federal Agency); 359th Medical Operations Squadron (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Jeffrey A. Cigrang, Dr. Jeffrey A. Cigrang, Wright State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWH20150096H; W81XWH-15-2-0025 (Other Grant/Funding Number: USA Med Research ACQ Activity)
Record Dates: First submitted 2015-10-04; First posted 2015-10-08 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Marriage
Keywords: Military Couples; Marriage; Primary Care; Marriage Intervention; Air Force

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 7-Month Wait List Group (Experimental): Couples will be randomly assigned to a wait list group. This group will wait seven months before starting The Marriage Checkup.
  Interventions: Behavioral: Marriage Checkup
- MC Right Away (Experimental): Couples will be randomly assigned to receive The Marriage Checkup right away.
  Interventions: Behavioral: Marriage Checkup

INTERVENTIONS:
Behavioral: Marriage Checkup — The MC adapted for primary care consists of three 30-minute appointments with the IBHC. Session 1 consists of discussing the of the couple's relationship history and each partner's primary strengths. Session 2 focuses on each partner's primary concern about the relationship. Session 3 is dedicated to providing feedback for the couple that identifies strengths, areas for possible improvement, and a menu of possible strategies or resources for the couple to consider pursuing.

SUMMARY:
The psychological health of military members is a critical element of force health protection and readiness. Frequent deployments and high operations tempo at home strain the relationships and families of today's military more than ever before (e.g., Karney & Crown, 2007). Since 2001 the likelihood of divorce in the Air Force increased with the number of days that Airmen were deployed (Karney & Crown, 2007). Distressed relationships not only adversely affect members' adjustment and readiness (e.g., Hoge et al., 2006) but also are centrally implicated in suicides (i.e., relationship problems are the precipitating event in 51% of Air Force suicides, Kindt, 2009) and domestic violence (Pan, Neidig, & O'Leary, 1994). Unfortunately, traditional sources of marriage counseling available to service members are largely underutilized. The MC brings a fresh perspective that helps normalize relationship help-seeking and in turn reach larger numbers of distressed couples early. The partnering of MC and integrated primary care appears to be an ideal combination of behavioral health innovations that has the potential to measurably enhance relationship health for the military services.

DETAILED DESCRIPTION:
The most challenging community problems faced by senior military leaders are closely linked to the quality of marriage relationships. These include family violence, spouse maltreatment, and suicide. Half (51%) of the service members who either completed or attempted suicide from 2008 to 2010 had a history of a failed intimate relationship, and for nearly one-third (30%) this failure had occurred within 30 days of the self-harm event. Relationship distress not only affects marriages but is also associated with depression, substance abuse, work role impairment and lowered children's health. Despite the potential high costs of chronic marital distress, very few couples seek therapy. In a recent Air Force study, only 6% of Airmen in distressed relationships reported making use of couple counseling after returning from deployment. Indeed, distressed couples wait an average of 6 years before seeking help, at which point their relationship likely has deteriorated dramatically.

Thus, there is a substantial need in the military for early detection and preventative care for deteriorating couples before serious and irreversible relationship damage has occurred. There are currently no widely available means to fill this need. Mild-to-moderately distressed couples may view therapy as reserved for only the most severely distressed couples, and thus delay seeking treatment until its efficacy is seriously diminished by the chronicity and severity of the accumulated relationship dysfunction.

The Marriage Checkup (MC) addresses this issue by providing a less-threatening option for couples to seek early preventative care before they have begun to identify as distressed. Intended to be the relationship health equivalent of the annual physical or dental checkup, the MC is a 4 to 5 hour assessment and feedback intervention. This brief intervention includes assessment of the couple's relationship history, strengths, and concerns and provides individualized feedback to the couple with a list of options addressing the couple's primary concerns. Studies conducted with civilian samples have shown that couples receiving MC demonstrate significant and lasting improvement across a range of marital health variables. In addition, MC has been shown to attract couples across the distress continuum and be perceived by couples as more accessible than traditional therapy.

In recognition of the limited reach and potential stigma of tertiary mental health treatment, the military services and the Department of Veterans Affairs have implemented collaborative care models in primary care. In a collaborative care model, mental health providers are embedded into the primary care setting and serve as integrated behavioral health consultants (IBHCs) to the medical providers. The IBHC provides brief, focused assessments and interventions for patients referred by their primary care provider. Marital problems are a common reason for primary care providers to refer patients to IBHCs, yet there has been no effort toward development of marital interventions suitable for primary care. MC's design as a brief "check-up" model for marriage help appeared particularly well-suited to primary care. Therefore, the investigators conducted a pilot study to adapt MC for use with military couples in Air Force primary care clinics (FWR20120054H).

In our pilot study the original MC was adapted for military couples and fit into the fast-paced environment of primary care. Military specific content for the assessment tools in the Marriage Checkup were developed. In addition, the team developed and piloted a protocol to use when only one member of the couple is available to come in for a Marriage Checkup, given the likelihood that some partners seeking an MC may have a partner who is currently deployed or otherwise unable/unwilling to participate in an in-person checkup. Finally, the Marriage Checkup was streamlined to fit within a Primary Care setting. More specifically, it was re-formatted into three 30-minute sessions. Session 1 consisted of the couple's relationship history and each partner's primary strengths, Session 2 focused on each partner's primary concern, and Session 3 is dedicated to feedback for the couple. IBHCs working in primary care were then trained to offer the intervention within a quasi-experimental research design in which pre-post changes were evaluated within subjects.

To date, twenty-two couples and one individual (N = 45; at least one partner in each couple was active duty) at two primary care sites have completed the MC. A multilevel modeling analysis indicated statistically significant pre-post changes for all study variables at both two weeks and two months, with effect sizes in the moderate range. Relationship satisfaction (B = .54, p = .003, B = .55, p = .004), distress (B = .75, p < .001, B = .58, p = .003) and intimacy (B = .43, p < .017, B = .47, p = .014) were significantly improved. In addition, couples completed a questionnaire measuring their level of satisfaction with the MC intervention itself. The scale ranged from 1(not at all) to 5 (very much), and across the questions the average response was 4.33 immediately post checkup and 4.05 at the one-month follow-up, indicating that couples were satisfied with their Marriage Checkup experience. The results of the pilot study provide preliminary evidence suggesting that the MC can be effectively adapted to a military population, and successfully used by behavioral health consultants (BHCs) working in an integrated primary care clinic.

The overall purpose of the proposed study is to build on pilot study findings by conducting a randomized trial of the military-adapted Marriage Checkup (MC) delivered in primary care by Integrated Behavioral Health Consultants (IBHCs). The primary outcomes of interest are marriage health (e.g., greater satisfaction, deeper intimacy) and community reach (e.g., attracts couples at-risk for marital deterioration who otherwise would not be seeking treatment). There are three specific objectives of the study, the first being to conduct a randomized trial comparing MC for use in military primary care clinics to a wait list control condition. Second, examine the effects of MC participation on relationship health at one month and six months post-treatment follow-up. Lastly, to determine whether the MC is successful at reaching couples at risk for marital deterioration who would otherwise be unlikely to seek traditional couple counseling.

This study will investigate two research hypotheses. The first hypothesis being that Military couples who participate in the Marriage Checkup (MC) for primary care will demonstrate positive relationship health trajectories for intimacy, acceptance, and relationship satisfaction over the course of six months when compared to couples in a wait-list control condition. A randomized control trial with 215 civilian couples demonstrated significant increases in relationship satisfaction, intimacy, and acceptance both in the short term and at two-year follow-up for treatment couples compared to no-treatment control couples. Emerging evidence further suggests that the primary mediator of improvements in marital health is the effect of the MC on increasing the level of intimate connection between spouses. In addition, the MC worked to affect both distal (i.e., depression) and specific (i.e., time together, sexual satisfaction and communication) outcomes. The second hypothesis is that the MC will attract military couples at-risk for marital deterioration who are otherwise not seeking relationship treatment. The MC is designed to significantly lower the barriers to couple help seeking. The MC is very brief and is advertised as an informational marital health service rather than therapy, intended for all couples who are interested in learning more about their strengths and areas of concern. The MC has been shown to attract a broad range of couples across the range of satisfaction from relationally satisfied to severely distressed and has been shown to successfully attract couples who would not otherwise seek any kind of relationship intervention.

The randomized trial will be conducted at four military primary care clinics. Three sites will be Wilford Hall Ambulatory Services Center (WHASC) in San Antonio, Texas, 359th Medical Operations Squadron (359 MDOS) in San Antonio, Texas, and Malcolm Grow Medical Clinics and Surgery Center (MGMCSC), Joint Base Andrews, in Maryland. The remaining site will be recommended by the Air Force Chief of Behavioral Health Optimization (co-investigator Maj Liz Najera).

Individuals and couples who express an interest in participating in the study will be scheduled by the on-site study coordinator with the IBHC to receive a more thorough explanation of the study purpose and requirements of participation. Potential participants will have the opportunity to ask questions about the study prior to making a decision to participate. Potential participants will be told that the MC involves three appointments with the IBHC within a four week period and completion of take-home relationship questionnaires to aid the BHC in assessing their relationship. At the third IBHC appointment the participants will receive feedback on the clinical questionnaires and interview results and be given a list of possible strategies for improving their relationship that has been tailored to their unique situation. For the purposes of the research, potential participants will be informed that they will be contacted approximately one month and six months later and asked to log onto a study website to re-complete surveys about their relationship. They will also complete surveys that ask their opinion of the MC including what they thought was most helpful and how it could be improved further.

This first contact will also include the standard brief clinical screening conducted by the IBHC for all referrals. During this screening the IBHC will also assess for the presence of any study exclusion factors. If at the conclusion of this first IBHC contact the potential participant expresses interest in participating and meets the inclusion and exclusion criteria, they will then meet with the Research Assistant to review and complete the informed consent documents for study participation and the baseline questionnaires.

The study will use a randomized two-group research design in which participants are randomly assigned after signing the informed consent document to either receive the MC right away or be placed on a 7-month wait list condition. All participants will complete study measures at baseline, eight weeks (1 month post-treatment for those assigned first to the MC condition) and 28 weeks (six months post-treatment for those assigned first to the MC condition). Participants assigned to the 7-month wait-list condition will be offered the MC at the completion of the 6-month follow-up measures.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants will be active duty and/or their active duty or Department of Defense (DoD) beneficiary spouses (adults >= 18 years old) who present to the IBHC in primary care with relationship concerns or questions following referral from their primary care manager or in response to study advertisements. Potential participants will be eligible for enrollment whether both partners are participating in-person or only one partner. Study participants do not have to be married; enrollment is open to active duty or who are not married but in committed romantic partnerships

Exclusion Criteria:

* Exclusion criteria will mirror clinical practice for patients normally not seen in primary care behavioral health, i.e., patients greater than mild risk for self-harm, patients with current alcohol dependence, psychotic disorder, significant dissociative disorder, or moderate or severe brain injury. Civilians along with potential participants that cannot understand, speak or read English will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2016-02; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
The Intimate Safety Questionnaire (ISQ) change from before MC and after MC | Participants will complete this measure at study enrollment, immediately after completion of the three Marriage Checkup appointments, and at a one-month post-treatment follow-up period.
  The ISQ (Cordova, Gee & Warren, 2005) is a 28-item measure of the degree to which partners feel safe being vulnerable with each other across several different domains of the relationship (Emotional Safety, Sexual Safety, Safety Disagreeing, Safety Being Yourself, and Safety in Public). Sample items include: I feel comfortable telling my partner when I'm feeling sad, sex with my partner makes me feel uncomfortable, and when I am with my partner I feel safe and comfortable. Scores range from 0 (never) to 4 (always). Negatively worded items are reversed scored such that higher scores indicate higher levels of intimacy.
Responsive Attention Scale (RAS) | Participants will complete this measure at study enrollment, immediately after completion of the three Marriage Checkup appointments, and at a one-month post-treatment follow-up period.
  Responsive Attention Scale (RAS; Trillingsgaard, 2013) is a 12-item scale measuring partners' responses to various bids for attention. The scale was developed for the Danish application of the Marriage Checkup. Items are rated on a 1(very rarely) to 5(very often) likert scale. Sample items include "I receive a warm welcome from my partner when we meet at the end of the day," "my partner smiles or laughs if I try to show him/her something funny," and "my partner is present and attentive when we eat together." Internal reliability for this measure has been high, with aplhas of .81 for both men and women.
Partner Compassion Scale | Participants will complete this measure at study enrollment, immediately after completion of the three Marriage Checkup appointments, and at a one-month post-treatment follow-up period.
  Partner Compassion Scale (PCS; Gray, Cordova & Maher, 2015). The PCS is a 9-item scale of compassionate expressions demonstrated by partners. This measure was developed to measure the primary mechanism of compassionate understand within the Marriage Checkup. Items are rated on a 0 (never) to 4 (always) likert scale. Sample items include " when my partner sees that I am hurting, he/she tries to comfort me," "even when he/she is upset or angry, my partner tries to be careful with my feelings," and "even when we disagree, my partner can put him/herself in my shoes." Since this measure was designed for the current study, it has not yet been tested for consistency and reliability.
Communication Skills Test | Participants will complete this measure at study enrollment, immediately after completion of the three Marriage Checkup appointments, and at a one-month post-treatment follow-up period.
  Communication Skills Test (CST; Saiz & Jenkins, 1995). The CST is a 10-item scale measuring communication skills within intimate relationships. Items are rated on a 1(almost never) to 7 (almost always) likert scale. Sample items include "I interrupt my partner when we are arguing" and "when discussing issues, I summarize what my partner says in order to make sure I understand him/her. Studies support the general reliability and validity of this measure (Stanley et al., 2001; Stanley et al., 2005).
Center for Epidemiological Studies Depression Scale - Short | Participants will complete this measure at study enrollment, immediately after completion of the three Marriage Checkup appointments, and at a one-month post-treatment follow-up period.
  Center for Epidemiologic Studies Depression Scale - Short (CES-D 10; adapted from Radloff 1977). The CES-D 10 is a shortened version of the CESD -20 and has demonstrated consistency and reliability consistent with the CESD-20 (Andresen, 1994). The CESD measures symptoms of depression within the previous week and uses a scale from Rarely or none of the time (less than one day) to All of the time (5-7 days). Sample items include "I felt lonely," "my sleep was restless," and "I felt like I could not 'get going.'" The CES-D has demonstrated good internal reliability and consistence (Cronbach's α = .88) (Thomas et al, 2008).
Couples Satisfaction Index (CSI) | Participants will complete this measure at study enrollment, immediately after completion of the three Marriage Checkup appointments, and at a one-month post-treatment follow-up period.
  Couples Satisfaction Index (CSI; Funk & Rogge, 2007). The CSI is a self-report questionnaire that assesses relationship satisfaction. Items include "please indicate the degree of happiness, all things considered, of your relationship" which is rated on a scale from 1 (extremely unhappy) to 6 (perfect) and "in general, how satisfied are you with your relationship?" which is rated on a scale from 0 (not at all) to 5 (completely). These four items have been selected from a larger pool of items which together contribute information to the construct of relationship satisfaction with arguably more precision than commonly used measures like the 32-item Dyadic Adjustment Scale (Spanier, 1976). The CSI has demonstrated excellent internal consistency, Cronbach's α equal to .94, and strong convergent validity with existing measures of relationship satisfaction by showing strong correlations with such measures, intercorrelations equal to .87 with the 32-item DAS and .91 with the 4-item DAS.
The Intimate Safety Questionnaire (ISQ) | Participants will complete this measure at study enrollment, immediately after completion of the three Marriage Checkup appointments, and at a one-month post-treatment follow-up period.
  The ISQ (Cordova, Gee & Warren,, 2005) is a 28-item measure of the degree to which partners feel safe being vulnerable with each other across several different domains of the relationship. Sample items include: I feel comfortable telling my partner when I'm feeling sad, sex with my partner makes me feel uncomfortable, and when I am with my partner I feel safe and comfortable. Scores range from 0 (never) to 4 (always). Negatively worded items are reversed scored such that higher scores indicate higher levels of intimacy. Internal reliability has been found to be adequate with alphas of .84 and .92 for men and women, respectively, and test-retest reliabilities of r = .89 and r = .91 for men and women, respectively. In the most recent MC study, internal reliability was high (Cronbach's α = 0.91) (Cordova et.al, in progress).

SECONDARY OUTCOMES:
Reasons For Seeking Marriage Checkup (RFSMC) | Participants will complete this measure at study enrollment.
  The RFSMC is a 2-item measure asking participants why would like to get a MC and how they hope to benefit from a MC.
Marriage Checkup Evaluation- Couple (MC Eval) change from immediately after MC and one month after MC | Immediately after completion of the three Marriage Checkup appointments, and at a one-month post-treatment follow-up period.
  The MC Eval is an 8-item measure assessing the couple's satisfaction with their Marriage Checkup. Sample items on the MC Eval include: do you feel your Marriage Checkup was helpful, do you feel the Marriage Checkup captured your relationship overall, and would you recommend the Marriage Checkup to other couples. Scores range from 1 (not at all) to 5 (very much) with higher scores indicating greater satisfaction with the Marriage Checkup.
Seeking Marriage Counseling Questionnaire | Immediately after completion of the three Marriage Checkup appointments, and at a one-month post-treatment follow-up period.
  The Seeking Marriage Counseling Questionnaire is a 2-item measure at Baseline and a 2-item measure at Followup designed to assess if the couple has ever seeked marriage counseling and if they sought marriage counseling upon completing the MC. Items on the Seeking Marriage Counseling Questionnaire include: if The Marriage Checkup was not available to you in primary care, would you have sought marriage counseling services from somewhere else, have you ever sought any type of marriage counseling for your current relationship before, and have you sought any type of marriage counseling since completing your Marriage Checkup? Scores range from definitely not to definitely and include qualitative responses.
Home-Work Stress Spillover | Immediately after completion of the three Marriage Checkup appointments, and at a one-month post-treatment follow-up period.
  The Home-Work Stress Spillover is a 12-item measure of the amount to which partners feel their relationship stress impacts their work functioning. Sample items on the Home-Work Stress Spillover include: caused you to feel drained of energy needed for your work, caused you to make mistakes at work, and reduced your overall job performance. Score range from never to several times per week. The spillover scale was developed by Dilworth (2004) for a study of dual-career mothers and fathers. Internal consistency of the items used in the Dolworth (2004) study was good (Cronbach's alpha = .77).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Cigrang, Ph.D., Principal Investigator — Wright State University
Locations (2):
- United States (2):
  - Wright-Patterson Air Force Base, Fairborn, Ohio
  - Wilford Hall Ambulatory Surgical Center, San Antonio, Texas

REFERENCES:
- [Background] Bush NE, Reger MA, Luxton DD, Skopp NA, Kinn J, Smolenski D, Gahm GA. Suicides and suicide attempts in the U.S. Military, 2008-2010. Suicide Life Threat Behav. 2013 Jun;43(3):262-73. doi: 10.1111/sltb.12012. Epub 2013 Jan 17. PMID 23330611
- [Background] Cummings EM, Goeke-Morey MC, Papp LM. Children's responses to everyday marital conflict tactics in the home. Child Dev. 2003 Nov-Dec;74(6):1918-29. doi: 10.1046/j.1467-8624.2003.00646.x. PMID 14669904
- [Background] Gottman, J. M. & Gottman, J.S. (1999). The marriage survival kit. In R. Berger & M.T. Hannah (Eds.), Preventative approaches in couples therapy (pp 304-330). Philadelphia, PA: Brunner/Mazel.
- [Background] Cordova, J. V., Scott, R. L., Dorian, M., Mirgain, S., Yaeger, D., & Groot, A. (2005). The marriage checkup: A motivational interviewing approach to the promotion of marital health with couples at-risk for relationship deterioration. Behavior Therapy, 36, 301-310.
- [Background] Cordova JV, Fleming CJ, Morrill MI, Hawrilenko M, Sollenberger JW, Harp AG, Gray TD, Darling EV, Blair JM, Meade AE, Wachs K. The Marriage Checkup: a randomized controlled trial of annual relationship health checkups. J Consult Clin Psychol. 2014 Aug;82(4):592-604. doi: 10.1037/a0037097. Epub 2014 Jun 16. PMID 24932565
- [Background] Gee CB, Scott RL, Castellani AM, Cordova JV. Predicting 2-year marital satisfaction from partners' discussion of their marriage checkup. J Marital Fam Ther. 2002 Oct;28(4):399-407. doi: 10.1111/j.1752-0606.2002.tb00365.x. PMID 12382549
- [Background] Morrill MI, Eubanks-Fleming C, Harp AG, Sollenberger JW, Darling EV, Cordova JV. The marriage checkup: increasing access to marital health care. Fam Process. 2011 Dec;50(4):471-85. doi: 10.1111/j.1545-5300.2011.01372.x. PMID 22145720
- [Background] Maguen, S., Cohen, G., Cohen, B. E., Lawhon, G. D., Marmar, C. R., & Seal, K. H. (2010). The role of psychologists in the care of Iraq and Afghanistan veterans in primary care settings. Professional Psychology: Research and Practice, 41, 135-142.
- [Background] Gray, T.D, Hawrilenko, M.J., & Cordova, J.V. (in progress). Distal and Specific Outcomes of the Marriage Checkup.
- [Background] Karney, B. R., & Crown, J. S. (2007). Families under stress: An assessment of data, theory, and research on marriage and divorce in the military. Santa Monica, CA: RAND Corporation.
- [Background] Hoge CW, Auchterlonie JL, Milliken CS. Mental health problems, use of mental health services, and attrition from military service after returning from deployment to Iraq or Afghanistan. JAMA. 2006 Mar 1;295(9):1023-32. doi: 10.1001/jama.295.9.1023. PMID 16507803
- [Background] Kindt, M. (2009). Talking paper on 2008 AF suicide trends. Unpublished manuscript, AF Medical Operations Agency.
- [Background] Pan HS, Neidig PH, O'Leary KD. Predicting mild and severe husband-to-wife physical aggression. J Consult Clin Psychol. 1994 Oct;62(5):975-81. doi: 10.1037//0022-006x.62.5.975. PMID 7806729
- [Background] Whisman MA, Uebelacker LA. Impairment and distress associated with relationship discord in a national sample of married or cohabiting adults. J Fam Psychol. 2006 Sep;20(3):369-77. doi: 10.1037/0893-3200.20.3.369. PMID 16937993
- [Background] Wilson, P. G. (2003). The Air Force experience: Integrating behavioral health providers into primary care. In R. G. Frank, S. H. McDaniel, J. H. Bray, & M. Heldring (Eds.), Primary care psychology, Washington DC: American Psychological Association.
- [Background] Seal KH, Cohen G, Bertenthal D, Cohen BE, Maguen S, Daley A. Reducing barriers to mental health and social services for Iraq and Afghanistan veterans: outcomes of an integrated primary care clinic. J Gen Intern Med. 2011 Oct;26(10):1160-7. doi: 10.1007/s11606-011-1746-1. Epub 2011 Jun 7. PMID 21647750
- [Derived] Cigrang JA, Cordova JV, Gray TD, Fedynich AL, Maher E, Diehl AN, Hawrilenko M. Marriage checkup in integrated primary care: A randomized controlled trial with active-duty military couples. J Consult Clin Psychol. 2022 May;90(5):381-391. doi: 10.1037/ccp0000734. PMID 35604745